CLINICAL TRIAL: NCT03137381
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of CTP-543 in Adult Patients With Moderate to Severe Alopecia Areata
Brief Title: Study to Evaluate the Safety and Efficacy of CTP-543 in Adults With Moderate to Severe Alopecia Areata
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP543.2001
Record Dates: First submitted 2017-04-28; First posted 2017-05-02 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: CTP-543 4 mg BID (Experimental): Participants will receive CTP-543 4 mg tablets, twice daily for up to 24 weeks.
  Interventions: Drug: CTP-543
- Cohort 2: CTP-543 8 mg BID (Experimental): Participants will receive CTP-543 8 mg tablets, twice daily for up to 24 weeks.
  Interventions: Drug: CTP-543
- Cohort 3: CTP-543 12 mg BID (Experimental): Participants will receive CTP-543 12 mg tablets, twice daily for up to 24 weeks.
  Interventions: Drug: CTP-543
- Combined Placebo (Placebo Comparator): Participants will receive CTP-543 matched placebo tablets, twice daily for up to 24 weeks in Cohorts 1, 2, and 3.
  Interventions: Drug: CTP-543 matching placebo

INTERVENTIONS:
Drug: CTP-543 — Administered as tablets.
  Arms: Cohort 1: CTP-543 4 mg BID; Cohort 2: CTP-543 8 mg BID; Cohort 3: CTP-543 12 mg BID
Drug: CTP-543 matching placebo — Administered as tablets.
  Arms: Combined Placebo

SUMMARY:
This study will evaluate the safety and efficacy of CTP-543 on hair loss in adults with chronic, moderate to severe alopecia areata.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled multi-center study consisting of 3 cohorts to assess the safety and efficacy of CTP-543. Each Cohort will be initiated sequentially in ascending dose order. Participants will be randomized to either an active dose of CTP-543 or placebo for a 24-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of alopecia areata with a current episode lasting at least 6 months and not exceeding 10 years at the time of Screening. Total disease duration greater than 10 years is permitted.
* At least 50% scalp hair loss, as defined by a Severity of Alopecia Tool (SALT) score ≥50, at Screening and Baseline.
* Clinical lab results within the normal range

Exclusion Criteria:

* Active scalp inflammation, psoriasis, or seborrheic dermatitis requiring topical treatment to the scalp, significant trauma to the scalp, or untreated actinic keratosis on the scalp.
* Treatment with systemic immunosuppressive medications or biologics.
* Vaccination with herpes zoster vaccine or any live virus within 6 weeks of screening or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen E. Hamilton, Study Director — Concert Pharmaceuticals, Inc.
Locations (13):
- United States (13):
  - University of California, Irvine, Irvine, California
  - Contour Dermatology & Cosmetic Surgery Center, Rancho Mirage, California
  - Stanford University School of Medicine, Redwood City, California
  - Kaiser Permanente Northern California, San Francisco, California
  - Yale School of Medicine, New Haven, Connecticut
  - Siperstein Dermatology Group, Boynton Beach, Florida
  - Northwestern University, Chicago, Illinois
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Northwest Dermatology, Portland, Oregon
  - Suzanne Bruce & Associates, PA, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cassella J, Hamilton C, von Hehn J, Braman V. JAK Inhibitor CTP-543 Achieves Primary Endpoint in Phase 2 Trial in Alopecia Areata. In: Proceedings from the 2019 American Academy of Dermatology Meeting; 01-05 March 2019; Washington, DC. Abstract 11291.
- [Background] Cassella J, Hamilton C, von Hehn J, Braman V. JAK Inhibitor CTP-543 Achieves Primary Endpoint in Phase 2 Trial in Alopecia Areata. In: Proceedings from the 11th World Congress Hair Research; 24-27 April 2019; Sitges, Barcelona.
- [Background] Cassella J, Hamilton C, von Hehn J, Braman V. CTP-543, an oral JAK inhibitor, achieves primary endpoint in Phase 2 randomized, placebo-controlled, dose ranging trial in patients with moderate to severe alopecia areata. In: Proceedings from the 28th EADV Congress; 09-13 October 2019, Madrid, Spain. D3T01.1: Late breaking news.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 13 study centers in the United States from 09 August 2017 to 08 July 2019.
Pre-assignment Details: 235 participants were screened, out of which 149 participants who experienced an episode of hair loss due to alopecia areata were enrolled to receive CTP-543 or placebo.
Groups:
- Combined Placebo: Participants received CTP-543 matched placebo tablets, twice daily for up to 24 weeks in Cohorts 1, 2, and 3.
- Cohort 1: CTP-543 4 mg BID: Participants received CTP-543 4 mg tablets, twice daily for up to 24 weeks.
- Cohort 2: CTP-543 8 mg BID: Participants received CTP-543 8 mg tablets, twice daily for up to 24 weeks.
- Cohort 3: CTP-543 12 mg BID: Participants received CTP-543 12 mg tablets, twice daily for up to 24 weeks.
Period: Overall Study
Arm/Group | Combined Placebo | Cohort 1: CTP-543 4 mg BID | Cohort 2: CTP-543 8 mg BID | Cohort 3: CTP-543 12 mg BID
Started | 44 | 30 | 38 | 37
Safety Population (Safety Population included all participants who received study drug during the treatment period. Participants were analyzed according to the actual treatment received during the study.) | 44 | 29 | 38 | 36
Completed | 35 | 23 | 30 | 36
Not Completed | 9 | 7 | 8 | 1
Not completed — Adverse Event | 3 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0
Not completed — Protocol deviation | 1 | 1 | 0 | 1
Not completed — Withdrawal by Investigator | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 3 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population included all the randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Placebo | Cohort 1: CTP-543 4 mg BID | Cohort 2: CTP-543 8 mg BID | Cohort 3: CTP-543 12 mg BID | Total
Number analyzed (Participants) | 44 | 30 | 38 | 37 | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (13.50) | 35.7 (11.01) | 37.3 (14.18) | 35.8 (12.37) | 36.8 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 22 | 26 | 28 | 105
  Male | 15 | 8 | 12 | 9 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 4 | 3 | 15
  Not Hispanic or Latino | 39 | 26 | 33 | 34 | 132
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 7 | 2 | 7 | 3 | 19
  White | 33 | 25 | 26 | 30 | 114
  Other | 1 | 1 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving at Least a 50% Relative Reduction in Severity of Alopecia Tool (SALT) Score From Baseline at Week 24
Description: The SALT is a quantitative assessment of scalp hair loss. SALT scores range in severity from 0 (no hair loss) to a maximum of 100 (complete hair loss). Responders were defined as participants achieving at least a 50% relative reduction in SALT score from baseline at Week 24.
Time Frame: Week 24
Population: Efficacy Population included all participants who received study drug and had at least 1 post-treatment SALT assessment during the treatment period. Participants were analyzed according to their randomized treatment group.
Measure: Number; unit: Percentage of participants
Arm/Group | Combined Placebo | Cohort 1: CTP-543 4 mg BID | Cohort 2: CTP-543 8 mg BID | Cohort 3: CTP-543 12 mg BID
Number analyzed (Participants) | 43 | 28 | 38 | 36
Percentage of participants | 9.3 | 21.4 | 47.4 | 58.3
Statistical Analysis 1: Comparison: Combined Placebo vs Cohort 1: CTP-543 4 mg BID; Test type: Superiority; p = 0.177, Chi-squared
Statistical Analysis 2: Comparison: Combined Placebo vs Cohort 2: CTP-543 8 mg BID; Test type: Superiority; p < 0.001, Chi-squared
Statistical Analysis 3: Comparison: Combined Placebo vs Cohort 3: CTP-543 12 mg BID; Test type: Superiority; p < 0.001, Chi-squared

2. Primary Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event is any untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the patient's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a pre-existing condition) should be considered an adverse event. TEAE is defined as any adverse event that occurs after administration of the first dose of study drug.
Time Frame: From first dose of study drug up to safety follow up at Week 28
Population: Safety Population included all participants who received study drug during the treatment period. Participants were analyzed according to the actual treatment received during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Placebo | Cohort 1: CTP-543 4 mg BID | Cohort 2: CTP-543 8 mg BID | Cohort 3: CTP-543 12 mg BID
Number analyzed (Participants) | 44 | 29 | 38 | 36
Participants | 31 | 25 | 31 | 30

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to safety follow up at Week 28
Description: All-cause mortality, Serious and other adverse events are reported for the Safety Population, included all participants who received study drug during the treatment period. Participants were analyzed according to the actual treatment received during the study.
Arm/Group | Combined Placebo | Cohort 1: CTP-543 4 mg BID | Cohort 2: CTP-543 8 mg BID | Cohort 3: CTP-543 12 mg BID
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/29 | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/29 | 0/38 | 1/36
Other Adverse Events (participants affected / at risk) | 31/44 | 25/29 | 31/38 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Placebo (N=44) | Cohort 1: CTP-543 4 mg BID (N=29) | Cohort 2: CTP-543 8 mg BID (N=38) | Cohort 3: CTP-543 12 mg BID (N=36)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Placebo (N=44) | Cohort 1: CTP-543 4 mg BID (N=29) | Cohort 2: CTP-543 8 mg BID (N=38) | Cohort 3: CTP-543 12 mg BID (N=36)
Upper respiratory tract infection (Infections and infestations) | 7 | 2 | 2 | 7
Nasopharyngitis (Infections and infestations) | 1 | 3 | 3 | 9
Folliculitis (Infections and infestations) | 0 | 3 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 1 | 0 | 2
Body tinea (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 2 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 3 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 3 | 0
Low density lipoprotein increased (Investigations) | 0 | 0 | 4 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 3 | 0
Hemoglobin decreased (Investigations) | 0 | 1 | 2 | 0
Amylase increased (Investigations) | 0 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Hematocrit decreased (Investigations) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Headache (Nervous system disorders) | 4 | 5 | 10 | 7
Migraine (Nervous system disorders) | 1 | 0 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 6
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 2 | 2 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 3
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator wants to publish study data or results, the publication or presentation must be provided to Concert for review at least 60 days in advance. If Concert needs to file a patent application prior to publication, the publication can be delayed up to 90 days from Sponsor providing notice to the investigator of such need.

DOCUMENTS (2):
  • Study Protocol (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT03137381/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/81/NCT03137381/SAP_001.pdf